CLINICAL TRIAL: NCT02150057
Title: Efficacy of Medial Compartment Unloading Brace Use for Osteoarthritis of the the Knee: A Prospective Randomized Study
Brief Title: Efficacy Study of an Unloading Brace for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: BREG, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BREG72609
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: knee osteoarthritis unicompartmental unloading brace
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Subjects who meet the recruitment conditions will be prospectively randomized into one of two treatment groups for 6 month evaluation:
  1. Breg Fusion Osteoarthritis Knee Brace
  2. No brace group Both groups will be allowed to continue standard conservative treatment of osteoarthritis including anti-inflammatory medications, home exercises and joint supplements.
Who Masked: Care Provider
Masking Description: Two orthopedic surgeons will blindly grade the osteoarthritis and calculate the mechanical axis and knee angles. The two surgeons' measurements will be averaged. One surgeon's measurements will be repeated to determine intra-observer reliability.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): This group receives no experimental bracing intervention in the study.
- Experimental Group (Active Comparator): This group will receive the Breg Fusion Osteoarthritis Knee Unloading Brace to wear for a determined amount of time per study protocol for the treatment of osteoarthritis pain.
  Interventions: Device: Breg Fusion Unloading Brace

INTERVENTIONS:
Device: Breg Fusion Unloading Brace — This group is assigned to wear an unloading brace and report pain and quality of life by completion of a pain diary and related questionnaires.
  Other Names: Breg Fusion Osteoarthritis Knee Unloading Brace
  Arms: Experimental Group

SUMMARY:
Subjects with symptomatic unicompartmental osteoarthritis of the knee will be invited to participate in this randomized study. Subjects will be assigned to either a Fusion Osteoarthritis Knee Brace group, or a control group that does not wear a brace. It is hypothesized that use of the Fusion Osteoarthritis Knee Brace will have a better outcome on osteoarthritis knee pain and quality of life compared to those who do not receive bracing intervention.

DETAILED DESCRIPTION:
This investigation will recruit 72 subjects from the clinical population of the investigators with symptomatic unicompartmental osteoarthritis of the medial compartment of the knee who meet the inclusion criteria of the investigation. Subjects who meet the recruitment conditions will be prospectively randomized into one of two treatment groups for 6 month evaluation:

1. Fusion Osteoarthritis Knee Brace
2. No brace group

Inclusion Criteria:

* Age 30-80.
* History of medial unicompartmental knee pain > 3 months duration (medial compartment only).
* Narrowing of medial joint space < one half of lateral compartment
* Varus deformity no greater than 80
* Mild to moderate limitation in Activities of Daily Living (ADL's) and/or recreational activities.
* Must read and understand English language and demonstrate the ability and willingness to follow the protocol and complete the questionnaires and diaries.
* Manual dexterity sufficient to perform all tasks required of study participants.
* Willingness to wear the brace a minimum of 4 hours per day.

Exclusion Criteria:

* Arthritides other than osteoarthritis.
* Previous high tibial osteotomy of the affected knee.
* Previous surgery of affected knee other than diagnostic arthroscopy with joint debridement, soft tissue reconstruction, menisectomy.
* Fixed flexion deformities / limitations >10 degrees as compared to the contralateral limb.
* Flexion limitation > 20 degrees.
* Significant soft tissue compromise preventing long-term brace use.
* Peripheral vascular disease or other neurovascular complaints

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80.
* History of medial unicompartmental knee pain > 3 months duration (medial compartment only).
* Narrowing of medial joint space < one half of lateral compartment
* Varus deformity no greater than 80
* Mild to moderate limitation in Activities of Daily Living (ADL's) and/or recreational activities.
* Must read and understand English language and demonstrate the ability and willingness to follow the protocol and complete the questionnaires and diaries.
* Manual dexterity sufficient to perform all tasks required of study participants.
* Willingness to wear the brace a minimum of 4 hours per day.

Exclusion Criteria:

* Arthritides other than osteoarthritis.
* Previous high tibial osteotomy of the affected knee.
* Previous surgery of affected knee other than diagnostic arthroscopy with joint debridement, soft tissue reconstruction, menisectomy.
* Fixed flexion deformities / limitations >10 degrees as compared to the contralateral limb.
* Flexion limitation > 20 degrees.
* Significant soft tissue compromise preventing long-term brace use.
* Peripheral vascular disease or other neurovascular complaints.
* Leg-length discrepancy > 2cm.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Ostrander, MD, Principal Investigator — Andrews Institute for Orthopaedics & Sports Medicine
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham LS, Kelsey JL. Epidemiology of musculoskeletal impairments and associated disability. Am J Public Health. 1984 Jun;74(6):574-9. doi: 10.2105/ajph.74.6.574. PMID 6232862
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Lethbridge-Cejku M, Tobin JD, Scott WW Jr, Reichle R, Plato CC, Hochberg MC. The relationship of age and gender to prevalence and pattern of radiographic changes of osteoarthritis of the knee: data from Caucasian participants in the Baltimore Longitudinal Study of Aging. Aging (Milano). 1994 Oct;6(5):353-7. doi: 10.1007/BF03324264. PMID 7893781
- [Background] Gabriel SE, Crowson CS, Campion ME, O'Fallon WM. Direct medical costs unique to people with arthritis. J Rheumatol. 1997 Apr;24(4):719-25. PMID 9101508
- [Background] Gabriel SE, Crowson CS, O'Fallon WM. Costs of osteoarthritis: estimates from a geographically defined population. J Rheumatol Suppl. 1995 Feb;43:23-5. PMID 7752127
- [Background] Rao JK, Mihaliak K, Kroenke K, Bradley J, Tierney WM, Weinberger M. Use of complementary therapies for arthritis among patients of rheumatologists. Ann Intern Med. 1999 Sep 21;131(6):409-16. doi: 10.7326/0003-4819-131-6-199909210-00003. PMID 10498556
- [Background] Buckwalter JA, Stanish WD, Rosier RN, Schenck RC Jr, Dennis DA, Coutts RD. The increasing need for nonoperative treatment of patients with osteoarthritis. Clin Orthop Relat Res. 2001 Apr;(385):36-45. doi: 10.1097/00003086-200104000-00008. PMID 11302324
- [Background] Pollo FE. Bracing and heel wedging for unicompartmental osteoarthritis of the knee. Am J Knee Surg. 1998 Winter;11(1):47-50. No abstract available. PMID 9606092
- [Background] Pollo FE, Otis JC, Backus SI, Warren RF, Wickiewicz TL. Reduction of medial compartment loads with valgus bracing of the osteoarthritic knee. Am J Sports Med. 2002 May-Jun;30(3):414-21. doi: 10.1177/03635465020300031801. PMID 12016084
- [Background] Matsuno H, Kadowaki KM, Tsuji H. Generation II knee bracing for severe medial compartment osteoarthritis of the knee. Arch Phys Med Rehabil. 1997 Jul;78(7):745-9. doi: 10.1016/s0003-9993(97)90083-6. PMID 9228878
- [Background] Kirkley A, Webster-Bogaert S, Litchfield R, Amendola A, MacDonald S, McCalden R, Fowler P. The effect of bracing on varus gonarthrosis. J Bone Joint Surg Am. 1999 Apr;81(4):539-48. doi: 10.2106/00004623-199904000-00012. PMID 10225800
- [Background] Katsuragawa Y, Fukui N, Nakamura K. Change of bone mineral density with valgus knee bracing. Int Orthop. 1999;23(3):164-7. doi: 10.1007/s002640050337. PMID 10486029
- [Background] Giori NJ. Load-shifting brace treatment for osteoarthritis of the knee: a minimum 2 1/2-year follow-up study. J Rehabil Res Dev. 2004 Mar;41(2):187-94. doi: 10.1682/jrrd.2004.02.0187. PMID 15558372
- [Background] Draper ER, Cable JM, Sanchez-Ballester J, Hunt N, Robinson JR, Strachan RK. Improvement in function after valgus bracing of the knee. An analysis of gait symmetry. J Bone Joint Surg Br. 2000 Sep;82(7):1001-5. doi: 10.1302/0301-620x.82b7.10638. PMID 11041589
- [Background] Divine JG, Hewett TE. Valgus bracing for degenerative knee osteoarthritis: relieving pain, improving gait, and increasing activity. Phys Sportsmed. 2005 Feb;33(2):40-6. doi: 10.3810/psm.2005.02.48. PMID 20086350
- [Background] Birmingham TB, Kramer JF, Kirkley A, Inglis JT, Spaulding SJ, Vandervoort AA. Knee bracing for medial compartment osteoarthritis: effects on proprioception and postural control. Rheumatology (Oxford). 2001 Mar;40(3):285-9. doi: 10.1093/rheumatology/40.3.285. PMID 11285375
- [Background] Barnes CL, Cawley PW, Hederman B. Effect of CounterForce brace on symptomatic relief in a group of patients with symptomatic unicompartmental osteoarthritis: a prospective 2-year investigation. Am J Orthop (Belle Mead NJ). 2002 Jul;31(7):396-401. PMID 12180625

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: Breg Fusion Osteoarthritis knee unloading brace
  Fusion Osteoarthritis Knee Brace: This group is assigned to wear an unloading brace and report pain and quality of life by completion of a pain diary and related questionnaires.
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 25 | 26
Completed | 19 | 22
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Population: 25 patients were enrolled in the control group but only 19 completed the study. 26 patients were enrolled in the experimental group but only 22 completed the study.
Groups:
- Experimental Group: This group is assigned to wear the BREG Fusion Osteoarthritis Unloading Brace and report pain and quality of life by completion of a pain diary and related questionnaires.
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.13 (6.11) | 67.8 (9.68) | 65.9 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Score
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be administered to collect patient reported outcomes as they relate to pain, function, and quality of life. The pain scale range is 0-10 with lower scores indicating less pain.
Time Frame: Baseline, 6 month follow-up
Population: Only 19 patients in the control group completed the study. Only 22 patients in the experimental group completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 19 | 22
units on a scale
  Baseline Visit | 2.92 (0.57) | 2.86 (0.52)
  6 Month Visit | 3.03 (0.65) | 2.67 (0.76)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for the 6 month duration that they were enrolled in the study.
Description: Our definition of adverse event does not differ from the clinicaltrials.gov definition.
Groups:
- Experimental Group: Breg Fusion Osteoarthritis knee unloading brace
  Fusion OA Knee Brace: This group is assigned to wear an unloading brace and report pain and quality of life by completion of a pain diary and related questionnaires.
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/22
Other Adverse Events (participants affected / at risk) | 3/19 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=19) | Experimental Group (N=22)
SOB/A-Fib (Cardiac disorders) | 0 | 1
Shingles (Nervous system disorders) | 0 | 1 — Hospitalization for shingles
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=19) | Experimental Group (N=22)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) — Rash/blisters
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There was difficulty recruiting subjects for this study which lead to a small number of subjects analyzed. The results of this study should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No